CLINICAL TRIAL: NCT03428165
Title: Transfer of Frozen Embryos in NATural Cycle: Evaluation of Impact of Spontaneous Versus HCG-triggered Ovulation on Pregnancy Rate - Bicentric Prospective Open Randomized Controlled Trial
Brief Title: Transfer of Frozen Embryos in Natural Cycle: Evaluation of Impact of Spontaneous Versus HCG-triggered Ovulation on Pregnancy Rate
Acronym: TECNAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-02/SH-01; 2017-A02759-44 (Other: ANSM)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-06

CONDITIONS: in Vitro Fertilization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human chorionic gonadotropin (HCG) (Other): Ovulation triggered using HCG: choriogonadotropin alpha (Ovitrelle, Merck Serono), 250 μg/0.5ml
  Interventions: Other: HCG
- spontaneous (No Intervention)

INTERVENTIONS:
Other: HCG — 250 μg/0.5ml choriogonadotropine alpha, Ovitrelle, Merck Serono
  Arms: human chorionic gonadotropin (HCG)

SUMMARY:
The purpose of the study is to evaluated whether there is a difference in pregnancy rate when transferring frozen embryos between patietns having spontaneously ovulated versus those triggered to voulate with HCG.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is aged between 18 and 40
* Patient has regular cycles and classified as 'easy' for transfer of a frozen embryo at blastocyste stage (vitrification day 5)

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient using donated oocytes
* Necessity of pre-implantation diagnosis
* Patients with stage 3 or 4 endometriosis or adenomyosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate after transfer of frozen embryos at day 14 between groups | Day 14
  Yes/no; Blood ßHCG > 100UI/L

SECONDARY OUTCOMES:
Pregnancy rate at week 12 | Week 12
  Yes/no; ultrasound
Miscarriage rate within first 12 weeks | Week 12
  Yes/no; ultrasound
Live birth | At delivery, maximum week 42
  Yes/no
Pregnancy term | At delivery, maximum week 42
  Weeks
Birth weight | At delivery, maximum week 42
  Kg
Cancellation of transfer due to premature ovulation (progesterone >3ng/ml and/or Luteinizing hormone > 3-fold base level) | Day 0
  Yes/no
Number of visits for endometrial preparation until attaining LH peak | Day 0
  Number of visits

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Huberlant, Principal Investigator — CHU Nimes
Locations (2):
- France (2):
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nimes, Nîmes

REFERENCES:
- [Result] Ranisavljevic N, Bonneau M, Rougier N, Hamamah S, Anahory T, Serand C, Huberlant S. Ovulation trigger versus spontaneous luteinizing hormone surge on live birth rate after frozen embryo transfer in a natural cycle: a randomized controlled trial. Fertil Steril. 2025 Apr;123(4):718-720. doi: 10.1016/j.fertnstert.2024.10.021. Epub 2024 Oct 19. No abstract available. PMID 39433204